CLINICAL TRIAL: NCT04569578
Title: Increasing Children's Physical Activity by Policy (CAP): a Cluster Randomized Controlled Trial in the Stockholm Region Preschools
Brief Title: Increasing Children's Physical Activity by Policy (CAP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm County Council (Center of Epidemiology and Community Medicine) (Unknown)
Responsible Party: Principal Investigator, Daniel Berglind, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAP2020
Record Dates: First submitted 2020-09-16; First posted 2020-09-30 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Physical Activity; Sedentary Behavior
Keywords: physical activity; preschool; randomized; intervention; sleep; sedentary behavior; sick leave
MeSH Terms: conditions — Motor Activity; Sedentary Behavior | interventions — Policy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Policy (Experimental): The policy will be implemented on preschool level.
  Interventions: Other: Policy
- Regular practice (No Intervention): The control preschool will continue their regular practice.

INTERVENTIONS:
Other: Policy — The intervention will include:
  i. Formalized physical activity policies implemented in preschools including the following:
  1. A minimum of 3 hours of total daily outdoor time scheduled both in the morning and in the afternoon
  2. At least 10 minutes teacher-led active play per day
  3. A minimum of 1 weekly outdoor excursion
  4. Meet the children outdoors when they arrive at preschool and/or picked up by their parents
  5. Only use screen tablets and computers for educational teaching purposes
  6. Communicating to, and encouraging, the parents to actively transport their children to and from preschools
  ii. A study website with an activity bank also serving as a platform for inter-professional education that preschool teachers can share and communicate about engaging activities and experience
  iii. Weekly follow-up and feedback by web-based questionnaires
  Arms: Policy

SUMMARY:
Levels of physical activity (PA) and physical fitness in children are low and declining, both globally and in Sweden. Preschools are important settings with the potential to influence the majority (>93%) of Swedish children's PA behaviors in early stage of life (<5 years). Preschool policy is an organizational level factor associated with children's PA but the casual link remains unclear. A cluster randomized controlled trial will be conducted to explore the feasibility and effectiveness of implementing a policy package for children's PA levels and other relevant health indicators.

DETAILED DESCRIPTION:
The overarching aim of the proposed project is to examine the effects of implementing physical activity (PA) policies in preschools on PA and indicators of health in young children. The proposed project is a unique collaboration between the applicants and Stockholm stad which will result in PA policies, that will be implemented in all 658 public preschools within the Stockholm region, having the possibility to affect more than 38 000 children.

The current study is designed as a cluster randomized controlled trial with 2 conditions (intervention vs. control) and preschools serving as the unit of randomization. Measures of primary and secondary outcomes will be obtained at baseline and at 6-months on an individual level.

This study will provide robust evidence of the effect of structural changes, at the organizational level of preschools, on children's PA and indicators of health. Notably, such robust evidence is urgently warranted as Swedish preschool children's PA levels are low which will have long-lasting effects on their lives. Finally, as the intervention has been developed in co-creation with Stockholm stad it has the possibility to, if proven effective, be implemented rapidly within preschools.

ELIGIBILITY:
Inclusion Criteria:

On preschool level:

* Located in Stockholm county
* Public preschool
* At least 60 children enrolled in preschool
* Chief of the preschool accepted the invitation for participation

On individual level-preschool children

* Enrolled in participating preschool
* 3-5 years old at the time of study start
* Parents signed informed consent
* Can participate in regular physical activity

On individual level-preschool teachers

* Full-time employee at the participating preschool
* Teachers responsible for participating children

Exclusion Criteria:

On preschool level:

* Located outside Stockholm county
* Private preschool
* Less than 60 children enrolled in preschool
* Chief of the preschool not willing to participate

On individual level-preschool children

* Not enrolled in participating preschool
* Outside 3-5 years old age range at study start
* Parents declined informed consent
* Cannot participate in regular physical activity due to mobility disability etc.

On individual level-preschool teachers

* Not full-time employee at the participating preschool
* Not responsible for any participating children

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4000 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity levels of children | Change from baseline 6 months follow-up in physical activity levels (daily minutes in moderate to vigorous physical activity)
  Physical activity levels in terms of daily minutes in moderate to vigorous physical activity, total physical activity and daily steps measured objectively by Actigraph GT3X+ accelerometers

SECONDARY OUTCOMES:
Change in sedentary time of children | Change from baseline to 6 months follow-up in daily minutes in sedentary time
  Daily sedentary time in minutes assessed by the Actigraph GT3X+
Change in musculoskeletal fitness of children | Change from baseline to 6 months follow-up in musculoskeletal fitness (handgrip strength)
  Musculoskeletal fitness, in terms of handgrip strength ,will be measured by an analogue dynamometer (TKK 5825, Grip-A, Takei, Tokyo, Japan).
Change in anthropometry (weight in kg) of children | Change from baseline to 6 months follow-up in anthropometry
  Weight will be measured by validated scales (calibrated scale: VB2-200-EC, Vetek AB, Väddö, Sweden)
Change in anthropometry (height in cm) of children | Change from baseline to 6 months follow-up in anthropometry
  Height will be measured by validated scales (portable stadiometer: Seca 213, Seca, Chino, CA, USA)
Change in anthropometry (waist circumference in cm) of children | Change from baseline to 6 months follow-up in anthropometry
  Waist circumference will be measured at the level of the navel directly on the skin
Change in anthropometry (BMI) of children | Change from baseline to 6 months follow-up in anthropometry
  Weight and height will be combined to report BMI in kg/m^2
Change in psychosocial functioning of children | Change from baseline to 6 months follow-up in psychosocial functioning
  Psychosocial functioning of children will be assessed by a parental proxy report of the Strength and Difficulty Questionnaire. Total difficulties score is generated by summing scores from all the scales except the prosocial scale and ranges from 0 to 40, higher score means worse outcome.
Change in sleep of children | Change from baseline to 6 months follow-up in sleep
  Sleep will be measured objectively by the GT3X+ accelerometer combined with a sleep time diary documented by parents during the days when the child is wearing the accelerometer. In addition, parents will answer questions about children's sleep duration and quality in the last 6 months in the sleep questionnaire. These sleep questions are adapted from the validated Ages and Stages Questionnaire. The sleep quality score ranges from 0-12 and higher score means better outcome.
Sick leave duration of children | From 12 months prior the intervention starts and during the 6 months intervention period
  Sick leave duration in terms of total days of leave will be collected from the Stockholm City smartphone application "Anmäl frånvaro".
Sick leave frequency of children | From 12 months prior the intervention starts and during the 6 months intervention period
  Sick leave frequency in terms of total occasions of leave will be collected from the Stockholm City smartphone application "Anmäl frånvaro".
Change in compliance with the World Health Organization (WHO) guidelines on physical activity, sedentary behaviour and sleep for children under 5 years of age | Change from baseline to 6 months follow-up in compliance with The WHO guidelines.
  World Health Organization (WHO) has published guidelines recommending more than 180 minutes of total physical activity with at least 60 minutes of moderate to vigorous physical activity, less than one hour of screen time and 10-13 hours of sleep across 24 hours
Change in physical activity levels of teachers | Change from baseline to 6 months follow-up in physical activity levels
  Physical activity levels in terms of daily minutes in moderate to vigorous physical activity measured by Actigraph GT3X+
Change in steps of teachers | Change from baseline to 6 months follow-up in steps
  Steps measured by Actigraph GT3X+
Change in sedentary time of teachers | Change from baseline to 6 months follow-up in daily minutes in sedentary time
  Daily sedentary time in minutes assessed by the Actigraph GT3X+
Change in musculoskeletal fitness of teachers | Change from baseline to 6 months follow-up in musculoskeletal fitness (handgrip strength)
  Musculoskeletal fitness, in terms of handgrip strength ,will be measured by an analogue dynamometer (TKK 5825, Grip-A, Takei, Tokyo, Japan).
Change in anthropometry (weight in kg) of teachers | Change from baseline to 6 months follow-up in anthropometry
  Weight validated scales (calibrated scale: VB2-200-EC, Vetek AB, Väddö, Sweden)
Change in anthropometry (height in cm) of teachers | Change from baseline to 6 months follow-up in anthropometry
  Height will be measured by validated scales (portable stadiometer: Seca 213, Seca, Chino, CA, USA)
Change in anthropometry (waist circumference in cm) of teachers | Change from baseline to 6 months follow-up in anthropometry
  Waist circumference will be measured at the level of the navel directly on the skin
Change in anthropometry (BMI) of teachers | Change from baseline to 6 months follow-up in anthropometry
  Weight and height will be combined to report BMI in kg/m^2
Sick leave duration of teachers | From 12 months prior the intervention starts and during the 6 months intervention period
  Sick leave duration in terms of total days of leave will be collected from the Stockholm City smartphone application "Anmäl frånvaro".
Sick leave frequency of teachers | From 12 months prior the intervention starts and during the 6 months intervention period
  Sick leave frequency in terms of total occasions of leave will be collected from the Stockholm City smartphone application "Anmäl frånvaro".

OTHER OUTCOMES:
Change in preschool policy and environmental characteristics (process outcome) | Change from baseline preschool policy and environmental characteristics at 3 months and at 6 months
  Preschool environmental characteristic such as available paly equipment, playground characteristic, policy, working practices will be assessed by validated Environment and Policy Evaluation and Observation as a Self-Report Instrument (EPAO-SR). The preschool playground characteristics and size will be double checked using google maps.
Implementation of the policy package (process outcome) | Measured weekly throughout 6 months only in intervention preschools
  Fidelity and dose of the implementation of the policy package will be documented through weekly feedback questionnaires throughout the intervention.
Normalization of the policy package into preschool teachers' regular practice (process outcome) | Measured at 6 months only in intervention preschools
  The extent to which the intervention can be normalized into preschool staff's regular practice will be assessed through No-MAD: Implementation measure based on Normalization Process Theory.
Change in children's physical activity opportunities outside preschool time (process outcome) | Change from baseline to 6 months follow-up in children's physical activity opportunities outside preschool time
  Children's PA opportunities in terms of active transport and participation in organized sports will be assessed via a questionnaire (daily during the period that children are wearing the accelerometers) where parents answer time, duration and type of organized sports and mode of transportation to and from preschool. In addition, several parental practices (outdoor time during the weekend, parental perception of physical activity, parental physical activity, and active play with parents) which could potentially influence children daily physical activity levels will also be assessed by questionnaire.
Project evaluation from parents | Measured at 6 months (questionnaires and interviews)
  How parents perceive and evaluate the intervention measured through questionnaire and interview.
Project evaluation from preschool teachers | Measured at 6 months ((questionnaires and interviews)
  How preschool teachers perceive and evaluate the intervention measured through questionnaire and interview.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Berglind, Associate Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen C, Ahlqvist VH, Henriksson P, Migueles JH, Christiansen F, Galanti MR, Berglind D. Increasing Children's physical Activity by Policy (CAP) in preschools within the Stockholm region: study protocol for a pragmatic cluster-randomized controlled trial. Trials. 2022 Jul 19;23(1):577. doi: 10.1186/s13063-022-06513-4. PMID 35854370
- See also: Project webside — https://ces.sll.se/var-verksamhet/aktiviteter-och-projekt/rorelseprojektet/